CLINICAL TRIAL: NCT05520099
Title: Observational Basket Trial to Collect Tissue to Develop and Train a Live Tumor Diagnostic Platform (ELEPHAS-02)
Brief Title: Observational Basket Trial to Collect Tissue to Develop and Train a Live Tumor Diagnostic Platform
Acronym: ELEPHAS-02
Status: Recruiting | Type: Observational
Sponsor: Elephas (Industry)
Responsible Party: Sponsor
Other Study IDs: ELEPHAS-02
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Immunotherapy; Cancer; Bladder Cancer; Urothelial Carcinoma Bladder; Kidney Cancer; Clear Cell Renal Cell Cancer (ccRCC); Colorectal Cancer; MSI-H Colorectal Cancer; DMMR Colorectal Cancer; Head and Neck Cancer (H&N); Squamous Cell Carcinoma Head and Neck Cancer (HNSCC); Liver Cancer; Hepatocellular Carcinoma (HCC); Lung Cancer (NSCLC); NSCLC (Non-small Cell Lung Cancer); Skin Cancer; Cutaneous Melanoma; Endometrial Cancer; Solid Tumor Cancer
Keywords: Immunotherapy; Live Tumor Fragment; Elephas; Elephas Score; Core Needle Biopsy; Forceps Biopsy; Punch Biopsy; Immune Checkpoint Inhibitors; Ex vivo Platform
MeSH Terms: conditions — Neoplasms; Urinary Bladder Neoplasms; Kidney Neoplasms; Carcinoma, Renal Cell; Colorectal Neoplasms; Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Liver Neoplasms; Carcinoma, Hepatocellular; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Skin Neoplasms; Melanoma; Endometrial Neoplasms | interventions — Biopsy, Large-Core Needle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh tissue sample using core needle biopsy, forceps biopsy, or punch biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected or diagnosed cancer types as listed in the description: Subjects suspected or diagnosed with recurrent, locally advanced or metastatic cancer: bladder (urothelial carcinoma), kidney (ccRCC).
  Subjects suspected or diagnosed with recurrent or metastatic cancer: Colon and Rectum (MSI-H/dMMR Colorectal Cancer), Head and Neck (Squamous Cell Carcinoma), liver (Hepatocellular Carcinoma), Lung (NSCLC), Skin (Cutaneous Melanoma), Uterus (endometrial cancer).
  Subjects suspected or diagnosed with one of the following cancer types eligible for pure ICI neoadjuvant therapy: Skin (Cutaneous Melanoma, Stage III)
  Subjects suspected or diagnosed with: Any solid tumor type that is eligible for pure ICI therapy in the neoadjuvant or advanced/metastatic setting; Any metastatic solid tumor with high TMB, MSI-High or dMMR and are being considered for treatment with ICI therapy; Any recurrent or metastatic patient with a solid tumor that the clinician plans to treat with ICI therapy.
  Interventions: Procedure: Core Needle Biopsy, Forceps Biopsy, Punch Biopsy

INTERVENTIONS:
Procedure: Core Needle Biopsy, Forceps Biopsy, Punch Biopsy — Subjects must be clinically able, at investigator discretion, to undergo additional core needle biopsy, forceps biopsy, or punch biopsy passes during their biopsy. These additional biopsies may either be collected from the primary tumor or a metastatic site amenable to additional passes (e.g., liver or lymph nodes) per the clinician.

SUMMARY:
The primary objective of this study is to develop and train the Elephas live tumor diagnostic platform and determine the ex-vivo accuracy of the Elephas Score using in-vivo RECIST 1.1 as the reference method

DETAILED DESCRIPTION:
Cancer is a leading cause of death and despite many new drugs, a major diagnostic challenge remains knowing which drug will work best for a patient. A new class of drugs called checkpoint inhibitors (CPIs) have revolutionized cancer treatment. However, current diagnostic methods (e.g. PDL1, MSI and TMB) do not accurately predict which patients will respond.

Elephas is developing a diagnostic platform using small 3D Live Tumor Fragments (LTFs) from participants for accurate prediction of drug response with a focus on CPIs such as Pembrolizumab (Keytruda). These LTFs contain both tumor cells and infiltrating immune cells, which are critical in determining response to CPIs and other immunotherapies.

In this observational clinical basket trial, participants will be recruited and their actual clinical response (using RECIST 1.1) to CPIs across five solid tumors (lung, head/neck, bladder, kidney, and skin) will be compared to the platform's predictive Artificial Intelligence (AI) score that is based on RNA, clinical data, and 3D microscopy images. The sensitivity and specificity of the platform's score will be determined and compared to current diagnostic methods for CPIs like PDL1, MSI, and TMB.

ELIGIBILITY:
Inclusion Criteria --

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. Subjects must meet one of the following criteria:

   * Subjects suspected or diagnosed with recurrent, locally advanced or metastatic cancer:

     * Bladder: Urothelial Carcinoma (UC)
     * Kidney: Clear Cell Renal Cell Carcinoma (ccRCC)
   * Subjects suspected or diagnosed with recurrent or metastatic cancer:

     * Colon and Rectum: Microsatellite instability-high (MSI-H)/deficient mismatch repair (dMMR) Colorectal Cancer (CRC)
     * Head and Neck: Squamous Cell Carcinoma (HNSCC), excluding nasopharyngeal and salivary gland cancers
     * Liver: Hepatocellular Carcinoma
     * Lung: Non-small cell lung cancer (NSCLC)
     * Skin: Cutaneous Melanoma, excluding Uveal Melanoma
     * Uterus: endometrial cancer
   * Subjects suspected or diagnosed with one of the following cancer types eligible for pure ICI neoadjuvant therapy:

     o Skin: Cutaneous Melanoma, Stage III
   * Subjects suspected or diagnosed with:

     * Any solid tumor type that is eligible for pure ICI therapy in the neoadjuvant or advanced/metastatic setting
     * Any metastatic solid tumor with high TMB, MSI-High or dMMR and are being considered for treatment with ICI therapy.
     * Any recurrent or metastatic patient with a solid tumor that the clinician plans to treat with ICI therapy.
4. Subjects must be clinically able, at investigator discretion, to undergo a biopsy procedure
5. Subjects who are newly diagnosed or have suspected cancer must be treatment-naïve at the time of biopsy. All other subjects should have the biopsy performed before starting their next line of treatment.

Exclusion Criteria --

1. Subjects who are pregnant
2. Subjects with a known auto-immune disease that would render them ineligible for immune-oncology treatment
3. Immunocompromised subjects, and subjects known to be HIV positive and currently receiving antiretroviral therapy
4. Subjects who are enrolled or plan to be enrolled in a blinded oncology treatment trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years or older, able to provide informed consent, and have a suspected or confirmed cancer diagnosis that meets requirements outlined in the eligibility criteria above.
Sampling Method: Non-Probability Sample
Enrollment: 416 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Determine Ex-Vivo Prognostic Accuracy of Elephas Platform | 3 years
  The ex-vivo prognostic accuracy of the Elephas live tumor diagnostic platform will be determined using in-vivo RECIST 1.1 as the reference method.

SECONDARY OUTCOMES:
Establish AUC of ELEPHAS Score and Compare with FDA Approved Biomarkers | 3 years
  The AUC of ELEPHAS Score will be established with a clinically meaningful confidence interval and compared to the AUCs of established FDA approved biomarkers for predicting clinical response to ICIs.

CONTACTS AND LOCATIONS:
Overall Officials: Fred Hausheer, MD, FACP, Study Director — Elephas
Locations (12):
- United States (12):
  - CARTI Cancer Center, Little Rock, Arkansas
  - Salinas Valley Memorial Healthcare System, Salinas, California
  - AdventHealth Orlando, Orlando, Florida
  - Memorial Health System, Pembroke Pines, Florida
  - Cleveland Clinic Florida, Stuart, Florida
  - University of South Florida (Tampa General Hospital), Tampa, Florida
  - University of Louisville James Graham Brown Cancer Center, Louisville, Kentucky
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen S, Zhang Z, Zheng X, Tao H, Zhang S, Ma J, Liu Z, Wang J, Qian Y, Cui P, Huang D, Huang Z, Wu Z, Hu Y. Response Efficacy of PD-1 and PD-L1 Inhibitors in Clinical Trials: A Systematic Review and Meta-Analysis. Front Oncol. 2021 Apr 16;11:562315. doi: 10.3389/fonc.2021.562315. eCollection 2021. PMID 33937012
- [Background] Cherukuri AR, Lubner MG, Zea R, Hinshaw JL, Lubner SJ, Matkowskyj KA, Foltz ML, Pickhardt PJ. Tissue sampling in the era of precision medicine: comparison of percutaneous biopsies performed for clinical trials or tumor genomics versus routine clinical care. Abdom Radiol (NY). 2019 Jun;44(6):2074-2080. doi: 10.1007/s00261-018-1702-1. PMID 30032384
- [Derived] Ramasubramanian TS, Adstamongkonkul P, Scribano CM, Johnson C, Caenepeel S, Hrycyniak LCF, Vedder L, Dana N, Baltes C, Browning T, Chen YI, Dietz T, Flietner E, Kaplewski N, Kellner A, Korrer M, Liu C, Marhefke N, McDonnell P, Nasreen A, Pope V, Prasad A, Richardson J, Schneider S, Schultz M, Sood C, Sunil A, von Euw E, Wait E, Wargowski E, Advani P, Broome B, Bruckbauer A, Godwin A, Kokabi N, Martin R, Robaina M, Toia G, Routh J, Friedl A, Eliceiri K, Szulczewski M, Johnson S, Oliner J, Galon J, Capitini C, Mukhopadhyay D, Taube J, Braun D, Gierman HJ. A live tumor fragment platform to assess immunotherapy response in core needle biopsies while addressing challenges of tumor heterogeneity. bioRxiv [Preprint]. 2025 Jul 18:2025.07.18.663728. doi: 10.1101/2025.07.18.663728. PMID 40791544